CLINICAL TRIAL: NCT06955052
Title: The Effects Of "Minds In Motion The Maze" on Balance and Gate In Children With Down Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/24/0746
Record Dates: First submitted 2025-04-24; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Down Syndrome
Keywords: Down syndrome; Minds in Motion; Cognitive behavior; Therapeutic approaches; Quality of life
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: The study will be randomized controlled trial. Total 20__ subjects will be assigned by non probability convenient sampling technique. They were randomly assigned to experimental and control groups. The Berg balance scale, limits of stability test, GOAL test, Timed up and go tools will be used. Tests will be used as outcome measure tools for balance, walk, coordination and Physical activity. All measures will be taken at baseline and at the end of treatment session. The collected data will be analyzed in Statistical Package for the Social Sciences (SPSS) 25.0 version. If data will be normally distributed then parametric if not normally distributed than non-parametric test will be apply.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group(MINDS IN MOTION THE MAZE) (Experimental): Clinical experimental: For group -mind in motion the maze at least for 7 weeks for 3 times per week during a period of 7 weeks intervention protocol : Balance board linear balance power skip jump rope tumble roll step ups midline touch
  Interventions: Other: "Minds In Motion The Maze"
- control group ( conventional treatment) (Active Comparator): Document any specific motor challenges or deficits typical in children with down syndrome.
  walk for 10 to 20 minutes warm up for 5 minutes cool down for 5 minutes rest period as per the subject convenience 6 stretching exercise performed during the warm and cool down period ,standing with feet together, standing with feet shoulder apart sitting with feet together ,sitting with feet shoulder width apart standing with only on leg extended , sitting with only one leg standing extended
  Interventions: Other: conventional treatment

INTERVENTIONS:
Other: "Minds In Motion The Maze" — "Minds in Motion the Maze" is a program that combines physical activity with cognitive training. Research suggests that MIM can positively impact balance and gait in children with Down syndrome. Some potential benefits include:
  * Improved balance and stability
  * Enhanced gross motor skills
  * Better coordination and overall physical function
  * Increased confidence in physical abilities
  The program's effectiveness may vary depending on individual needs and program implementation.
  Arms: experimental group(MINDS IN MOTION THE MAZE)
Other: conventional treatment — Document any specific motor challenges or deficits typical in children with down syndrome.
  walk for 10 to 20 minutes warm up for 5 minutes cool down for 5 minutes rest period as per the subject convenience 6 stretching exercise performed during the warm and cool down period ,standing with feet together, standing with feet shoulder apart sitting with feet together ,sitting with feet shoulder width apart standing with only on leg extended , sitting with only one leg standing extended
  Arms: control group ( conventional treatment)

SUMMARY:
This study explores the impact of "Minds In Motion: The Maze" on balance and gait in children with Down syndrome-a population often facing motor and coordination challenges. A randomized controlled trial will be conducted with 20 participants selected through non-probability convenience sampling and randomly assigned to experimental and control groups. The intervention group will engage in the "Minds In Motion: The Maze" program, designed to enhance motor skills through interactive activities. Balance and gait will be assessed using the Berg Balance Scale, Limits of Stability Test, GOAL Test, and Timed Up and Go test at baseline and post-intervention. Data will be analyzed using SPSS version 25.0, applying parametric or non-parametric tests based on distribution. Qualitative feedback from participants, parents, and instructors will also be gathered to assess the program's broader impact. This research aims to inform therapeutic strategies to improve motor function and independence in children with Down syndrome.

DETAILED DESCRIPTION:
This project aims to explore the effects of "Minds In Motion: The Maze" on the balance and gait of children diagnosed with Down syndrome. Down syndrome is a genetic disorder characterized by cognitive delays and physical challenges, including issues with balance and gait. "Minds In Motion: The Maze" is a specialized program designed to engage children in dynamic, interactive activities that target motor skills, coordination, and cognitive functions. The study will involve a sample of children diagnosed with Down syndrome, who will participate in the "Minds In Motion: The Maze" program for a specified duration. Their balance and gait will be assessed before and after the intervention using standardized tests and observational measures. Additionally, qualitative feedback from participants, parents, and instructors will be collected to gain insights into the perceived impact of the program. By investigating the effects of "Minds In Motion: The Maze" on balance and gait in children with Down syndrome, this research aims to contribute to the existing knowledge on interventions for enhancing motor skills and overall functioning in this population. The findings have the potential to inform the development of tailored therapeutic approaches to address the specific needs of children with Down syndrome, ultimately improving their quality of life and functional independence.

The study will be randomized controlled trial. Total 20__ subjects will be assigned by non probability convenient sampling technique. They were randomly assigned to experimental and control groups. The Berg balance scale, limits of stability test, GOAL test, Timed up and go tools will be used. Tests will be used as outcome measure tools for balance, walk, coordination and Physical activity. All measures will be taken at baseline and at the end of treatment session. The collected data will be analyzed in Statistical Package for the Social Sciences (SPSS) 25.0 version. If data will be normally distributed then parametric if not normally distributed than non-parametric test will be apply.

ELIGIBILITY:
Inclusion Criteria:

* Age group from 8 to 12 years
* Both male and female
* Children must have the physical and cognitive ability to engage in the activities
* Children should be in generally good health, without severe medical conditions or orthopedic issues
* Family consents

Exclusion Criteria:

* Uncontrolled seizures
* Any kind of orthopedic condition
* Registered visually impaired
* Atlanto Axial instability
* Any chest infection

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2025-06-05 (Estimated); Study Completion 2025-06-05 (Estimated)

PRIMARY OUTCOMES:
Balance berg scale | 7 weeks
  The Berg Balance Scale has been shown to have both high intra-rater and inter-rater reliability. Intra-rater reliability is when the same person who is administering the test can achieve the same results. Inter-rater reliability is when the test can be performed by different persons and achieve the same results. A systematic review conducted by Downs evaluated the Berg Balance Scale for individuals with various neurological conditions, including acute stroke, recent stroke, multiple sclerosis, cognitively impaired patients, and Parkinson disease patients, in different settings such as acute inpatient rehabilitation, outpatient rehabilitation, outpatient clinic, and home visits. The intra-rater relative reliability was found to be 0.98, with a 95% conference interval
Limits of stability test | 7 weeks
  Limits of Stability (LoS) is a significant variable in assessing stability and voluntary motor control in dynamic states. It provides valuable information by tracking the instantaneous change in the center of mass (COM) velocity and position. LoS is a useful measure for evaluating postural instability and identifying individuals at higher risk of falling, making it a valuable screening tool. Test-retest reliability ranged from high to low across the 5 LOS measures (intraclass correlation coefficient [2,k] = 0.82 to 0.48). Pearson correlations revealed 4 significant relationships (P < .05) between and within the 2 computerized posturography devices (r = 0.42 to -0.65)
GOAL Test | 7 weeks
  The Goal-Oriented Assessment of Life skills (GOAL) is an innovative new evaluation of functional motor abilities needed for daily living. Designed for children 7 to 17, the GOAL consists of seven Activities, fun and motivating tasks based on real occupations of a child's daily life. Each activity is linked to Intervention Targets that help you turn assessment results into a specific, goal-oriented treatment plan. This standardized, psycho metrically precise instrument offers an ecologically valid description of a child's competencies and opportunities for growth in both fine and gross motor domains.
Timed up and Go test | 7 weeks
  Timed Up and Go test (TUG) is a relatively simple test used to assess a person's mobility and requires both static and dynamic balance. The TUG is used frequently in the elderly population, as it is easy to administer and can generally be completed by most older adults has excellent inter-rater correlation (ICC) = 0.99, and high intra-rater reliability (ICC = 0.99

CONTACTS AND LOCATIONS:
Overall Officials: Wajeeha Saeed, MS-PPT, Principal Investigator — Riphah International University
Locations (1):
- Rising sun institute, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Terson de Paleville DGL, Immekus JC. A Randomized Study on the Effects of Minds in Motion and Yoga on Motor Proficiency and Academic Skills Among Elementary School Children. J Phys Act Health. 2020 Aug 15;17(9):907-914. doi: 10.1123/jpah.2019-0454. PMID 32805715